CLINICAL TRIAL: NCT03143777
Title: Does the Sara Combilizer®, an Early Mobilization Aid, Reduce the Time Taken to First Mobilise Ventilated Patients in Intensive Care?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David McWilliams, Clinical Specialist Physiotherapist, University Hospital Birmingham NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBirminghamNHS1
Record Dates: First submitted 2016-04-28; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Critical Illness
Keywords: physiotherapy; rehabilitation; critical care; seating
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Standard physiotherapy and mobilisation
- Sara Combilizer group (Experimental): Ongoing care with the sara combilizer available for use
  Interventions: Device: Sara Combilizer

INTERVENTIONS:
Device: Sara Combilizer — Combined tilt table and stretcher chair
  Arms: Sara Combilizer group

SUMMARY:
This study investigates the impact of introducing an early mobilisation device called the Sara Combilizer on time taken to mobilise in critical care. The investigators will collect baseline data on time taken to mobilise for a period of 4 months, then following a training programme and introduction of the device for a further 4 months

DETAILED DESCRIPTION:
Early mobility within the ICU is associated with a number of positive outcomes including reductions in ICU and hospital length of stay and better functional recovery. The exact definition of 'early' mobility is still not defined, with the actual ability to mobilize limited by a number of perceived factors.

The Sara Combilizer is a combined tilt table and stretcher chair, which allows passive transfer of patients out of bed. It is theorized the passive and safe nature of transfer may facilitate earlier mobilisation of patients within critical care. This study aimed to assess whether the introduction of the Sara Combilizer reduced time taken to first mobilize for patients mechanically ventilated for at least 5 days and at risk of ICU acquired weakness.

Patients admitted to a large UK critical care unit during the trial period and ventilated for ≥ 5 days were included in the study. Baseline data was collected prospectively for a period of 4 months. The Sara Combilizer was then introduced for a 1 month training and familiarization period, followed by a further 4 months prospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years) admitted to critical care and ventilated for 5 days or more

Exclusion Criteria:

* Patients with contraindications to mobilise (e.g. pelvic / spinal fractures)
* Poor prior level of mobility (<10yards)
* Neuromuscular disease (e.g. Guillain Barre or Motor Neurone Disease)
* Mechanical ventilation > 48 hours at another facility prior to admission
* Expected withdrawal of treatment within 24 next hours
* Patients who have already commenced mobilisation in the 1st 5 days of admission
* Obese patients who exceed the weight limit of the product (200 kg)
* Patients over 6ft5 due to restrictions of the product
* Severe neurological injury
* Lower limb amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time taken to 1st mobilise | Throughout ICU admission, average of 2 weeks
  Time taken to commence mobilisation , defined as sitting on the edge of the bed or out in a chair

SECONDARY OUTCOMES:
SOFA score | Throughout ICU admission, average of 2 weeks
  SOFA scores were calculated to measure degree of organ failure at the time of 1st mobilisation

IPD SHARING:
Plan to Share IPD: No